CLINICAL TRIAL: NCT02746393
Title: San Francisco General Hospital (SFGH) Health Advocates Phase II Study
Brief Title: SFGH Health Advocates Stage II Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 15-18305
Record Dates: First submitted 2015-12-01; First posted 2016-04-21 (Estimated); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Conditions Influencing Health Status; Social Determinants of Health

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Health Advocates Program
  Interventions: Other: Health Advocates Program
- 211 Arm (Active Comparator): 211 Information Sheet
  Interventions: Other: 211 Information Sheet

INTERVENTIONS:
Other: Health Advocates Program — Provided services and support to address identified social needs from health advocate navigators.
  Arms: Intervention
Other: 211 Information Sheet — Receive a printed list of community resources to address social needs.
  Arms: 211 Arm

SUMMARY:
The San Francisco General Hospital (SFGH) Health Advocate Staff II Study is a Randomized Controlled Trial (RCT) that collects survey data and non-invasive biological data from caregivers and children visiting a pediatric urgent care center. Families will be randomized according to a pre-determined randomization schedule into one of two social needs-focused interventions (the Health Advocates Program or a 211 Information active comparator arm). All patients in the study will be followed over a six month period to capture information about changes in social needs, health and health care utilization.

DETAILED DESCRIPTION:
Adverse social circumstances like hunger and food insecurity can have dramatic, negative impacts on the health of vulnerable children. In safety-net settings, the prevalence of these adverse social circumstances are high. The investigators are proposing an RCT on an intervention based in a large urban pediatric urgent care setting that addresses patients' social circumstances. In an earlier RCT conducted in a similar setting, this intervention helped decrease total social needs and parent reported child health on a single item measure. In this study, the investigators will collect a more robust set of survey data including detailed measures of child health and non-invasive biological data from children and caregivers accompanying those children. Families will be randomized according to a pre-determined randomization schedule into the social needs-focused intervention. In one arm, the investigators will offer the intervention, which involves in-person navigation around available social and legal resources; in the other, the investigators will offer written information to participants on available community resources. All patients in both arms will be followed over a six month period to capture information about changes in participants' social needs, health and health care utilization.

ELIGIBILITY:
Inclusion criteria:

* Child/Parent-Legal Guardian Caregiver Dyad;
* Child is SFGH Pediatric Urgent Care Clinic Patient between 0 and 17 years of age;
* Parent or Legal Guardian Caregiver over or equal to 18 years old;
* English or Spanish speaking Parent or Legal Guardian Caregiver;
* Both reside in San Francisco County.

Exclusion Criteria:

* Non-English or non-Spanish speaking Parent or Legal Guardian Caregiver;
* Parent or legal guardian caregiver under age 18;
* Parent or legal guardian caregiver accompanying patient is not familiar with the child's living situation;
* Family participated in study previously;
* Non-San Francisco County resident;
* Foster child or child in clinic for a child protective clearance exam.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1278 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Change in Caregiver Report of Child Health Status Using Pediatric Quality of Life Inventory (Peds QL) | Baseline and 6 months
  Collected at baseline and 6 month follow up
Change in Families' Social Needs Using Staff Administered Social Needs Screener | Baseline & 6 months
  Collected at baseline and 6 month follow up

SECONDARY OUTCOMES:
Change in caregiver depression using self-report PHQ | Baseline and 6 months
  measured at baseline and 6 months
Change in caregiver health using PROMIS-10 measures | Baseline and 6 months
  Collected at baseline and 6 month follow up
Change in Perceived Social Stress using self-report Perceived Stress Scale | Baseline and 6 Months
  Collected at baseline and 6 month follow up
Change in hair cortisol in children and caregivers | Baseline and 6 Months
  Collected at baseline and 6 month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Laura M Gottlieb, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Larson K, Halfon N. Family income gradients in the health and health care access of US children. Matern Child Health J. 2010 May;14(3):332-42. doi: 10.1007/s10995-009-0477-y. Epub 2009 Jun 5. PMID 19499315
- [Background] Wood PR, Smith LA, Romero D, Bradshaw P, Wise PH, Chavkin W. Relationships between welfare status, health insurance status, and health and medical care among children with asthma. Am J Public Health. 2002 Sep;92(9):1446-52. doi: 10.2105/ajph.92.9.1446. PMID 12197971
- [Background] Cook JT, Frank DA, Berkowitz C, Black MM, Casey PH, Cutts DB, Meyers AF, Zaldivar N, Skalicky A, Levenson S, Heeren T. Welfare reform and the health of young children: a sentinel survey in 6 US cities. Arch Pediatr Adolesc Med. 2002 Jul;156(7):678-84. doi: 10.1001/archpedi.156.7.678. PMID 12090835
- [Background] Frank DA, Neault NB, Skalicky A, Cook JT, Wilson JD, Levenson S, Meyers AF, Heeren T, Cutts DB, Casey PH, Black MM, Berkowitz C. Heat or eat: the Low Income Home Energy Assistance Program and nutritional and health risks among children less than 3 years of age. Pediatrics. 2006 Nov;118(5):e1293-302. doi: 10.1542/peds.2005-2943. PMID 17079530
- [Background] Meyers A, Cutts D, Frank DA, Levenson S, Skalicky A, Heeren T, Cook J, Berkowitz C, Black M, Casey P, Zaldivar N. Subsidized housing and children's nutritional status: data from a multisite surveillance study. Arch Pediatr Adolesc Med. 2005 Jun;159(6):551-6. doi: 10.1001/archpedi.159.6.551. PMID 15939854
- [Background] Garg A, Butz AM, Dworkin PH, Lewis RA, Serwint JR. Screening for basic social needs at a medical home for low-income children. Clin Pediatr (Phila). 2009 Jan;48(1):32-6. doi: 10.1177/0009922808320602. Epub 2008 Jun 19. PMID 18566347
- [Background] Lawton E, Leiter K, Todd J, Smith L. Welfare reform: advocacy and intervention in the health care setting. Public Health Rep. 1999 Nov-Dec;114(6):540-9. doi: 10.1093/phr/114.6.540. PMID 10670622
- [Background] Hanson M, Lawton E. Between a rock and a hard place: The prevalence and severity of unmet legal needs in the pediatric emergency department setting. Medical Legal Partnership for Children. 2007.
- [Background] Fleegler EW, Lieu TA, Wise PH, Muret-Wagstaff S. Families' health-related social problems and missed referral opportunities. Pediatrics. 2007 Jun;119(6):e1332-41. doi: 10.1542/peds.2006-1505. PMID 17545363
- [Background] Garg A, Butz AM, Dworkin PH, Lewis RA, Thompson RE, Serwint JR. Improving the management of family psychosocial problems at low-income children's well-child care visits: the WE CARE Project. Pediatrics. 2007 Sep;120(3):547-58. doi: 10.1542/peds.2007-0398. PMID 17766528
- [Background] Bikson K, McGuire J, Blue-Howells J, Seldin-Sommer L. Psychosocial problems in primary care: patient and provider perceptions. Soc Work Health Care. 2009;48(8):736-49. doi: 10.1080/00981380902929057. PMID 20182986
- [Background] Keller D, Jones N, Savageau JA, Cashman SB. Development of a brief questionnaire to identify families in need of legal advocacy to improve child health. Ambul Pediatr. 2008 Jul-Aug;8(4):266-9. doi: 10.1016/j.ambp.2008.04.004. Epub 2008 May 27. PMID 18644550
- [Background] Black MM, Cutts DB, Frank DA, Geppert J, Skalicky A, Levenson S, Casey PH, Berkowitz C, Zaldivar N, Cook JT, Meyers AF, Herren T; Children's Sentinel Nutritional Assessment Program Study Group. Special Supplemental Nutrition Program for Women, Infants, and Children participation and infants' growth and health: a multisite surveillance study. Pediatrics. 2004 Jul;114(1):169-76. doi: 10.1542/peds.114.1.169. PMID 15231924
- [Background] Jones SJ, Jahns L, Laraia BA, Haughton B. Lower risk of overweight in school-aged food insecure girls who participate in food assistance: results from the panel study of income dynamics child development supplement. Arch Pediatr Adolesc Med. 2003 Aug;157(8):780-4. doi: 10.1001/archpedi.157.8.780. PMID 12912784
- [Background] Cook JT, Frank DA, Berkowitz C, Black MM, Casey PH, Cutts DB, Meyers AF, Zaldivar N, Skalicky A, Levenson S, Heeren T, Nord M. Food insecurity is associated with adverse health outcomes among human infants and toddlers. J Nutr. 2004 Jun;134(6):1432-8. doi: 10.1093/jn/134.6.##. PMID 15173408
- [Background] Cook JT, Frank DA, Levenson SM, Neault NB, Heeren TC, Black MM, Berkowitz C, Casey PH, Meyers AF, Cutts DB, Chilton M. Child food insecurity increases risks posed by household food insecurity to young children's health. J Nutr. 2006 Apr;136(4):1073-6. doi: 10.1093/jn/136.4.1073. PMID 16549481
- [Background] Staufenbiel SM, Penninx BW, Spijker AT, Elzinga BM, van Rossum EF. Hair cortisol, stress exposure, and mental health in humans: a systematic review. Psychoneuroendocrinology. 2013 Aug;38(8):1220-35. doi: 10.1016/j.psyneuen.2012.11.015. Epub 2012 Dec 17. PMID 23253896
- [Background] Sharpley CF, McFarlane JR, Slominski A. Stress-linked cortisol concentrations in hair: what we know and what we need to know. Rev Neurosci. 2011 Dec 8;23(1):111-21. doi: 10.1515/RNS.2011.058. PMID 22150070
- [Background] Steptoe A, Hamer M, Chida Y. The effects of acute psychological stress on circulating inflammatory factors in humans: a review and meta-analysis. Brain Behav Immun. 2007 Oct;21(7):901-12. doi: 10.1016/j.bbi.2007.03.011. Epub 2007 May 1. PMID 17475444
- [Background] Weik U, Herforth A, Kolb-Bachofen V, Deinzer R. Acute stress induces proinflammatory signaling at chronic inflammation sites. Psychosom Med. 2008 Oct;70(8):906-12. doi: 10.1097/PSY.0b013e3181835bf3. Epub 2008 Sep 16. PMID 18799429
- [Background] Garg A, Toy S, Tripodis Y, Silverstein M, Freeman E. Addressing social determinants of health at well child care visits: a cluster RCT. Pediatrics. 2015 Feb;135(2):e296-304. doi: 10.1542/peds.2014-2888. Epub 2015 Jan 5. PMID 25560448
- [Derived] Pantell MS, Silveira PP, de Mendonca Filho EJ, Wing H, Brown EM, Keeton VF, Pokhvisneva I, O'Donnell KJ, Neuhaus J, Hessler D, Meaney MJ, Adler NE, Gottlieb LM. Associations between Social Adversity and Biomarkers of Inflammation, Stress, and Aging in Children. Pediatr Res. 2024 May;95(6):1553-1563. doi: 10.1038/s41390-023-02992-6. Epub 2024 Jan 17. PMID 38233512
- [Derived] Gottlieb LM, Adler NE, Wing H, Velazquez D, Keeton V, Romero A, Hernandez M, Munoz Vera A, Urrutia Caceres E, Arevalo C, Herrera P, Bernal Suarez M, Hessler D. Effects of In-Person Assistance vs Personalized Written Resources About Social Services on Household Social Risks and Child and Caregiver Health: A Randomized Clinical Trial. JAMA Netw Open. 2020 Mar 2;3(3):e200701. doi: 10.1001/jamanetworkopen.2020.0701. PMID 32154888